CLINICAL TRIAL: NCT01827618
Title: An Immunopharmacodynamic Phase 0/I Study of Rapamycin in Patients Undergoing Radical Cystectomy for Bladder Cancer
Brief Title: Neoadjuvant Rapamycin in Patients Undergoing Radical Cystectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Robert Svatek, Assistant Professor, Division of Urologic Oncology, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20120135H; KL2 TR000118-05/CTSA (Other: NIH/NCRR; UTHSCSA-Institute for Integration); KL2TR000118-05 (NIH)
Record Dates: First submitted 2013-03-29; First posted 2013-04-09 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Invasive Bladder Cancer Stage II
Keywords: bladder; Cancer; Cystectomy; Rapamycin
MeSH Terms: conditions — Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapamycin (Experimental): Rapamycin 3mg orally daily x 4weeks prior to radical cystectomy
  Interventions: Drug: Rapamycin
- Control (No Intervention)

INTERVENTIONS:
Drug: Rapamycin
  Other Names: Sirolimus, Rapamune
  Arms: Rapamycin

SUMMARY:
This study aims to evaluate the effects of rapamycin directly on bladder tumors and the effects of rapamycin on the immune system of patients with bladder cancer.

DETAILED DESCRIPTION:
This is a presurgical clinical trial which aims to understand the biologic activity of TORC1 inhibition and safety in patients with bladder cancer. In this presurgical setting, paired PMBCs and tumor tissue is evaluated before and after exposure to rapamycin to address target specificity, drug delivery, physiologic effects on tumor growth and apoptosis, and correlation of biomarkers with clinical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Have invasive (≥T1) bladder cancer
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. In their treating physician's opinion is a good candidate for radical cystectomy
4. In their treating physician's opinion does not need neoadjuvant chemotherapy prior to cystectomy
5. Be able to give informed consent
6. Be age 18 or older
7. Have adequate marrow function (defined as granulocytes greater than 1,500 cells/mm3 hemoglobin >9.5 gm/dl or platelets more than 100,000 cells/mm3).
8. Have adequate end-organ function (GFR >30, bilirubin <1.5, SGOT < 3x ULN)
9. Have a life expectancy > one year
10. Not have a prior history of non-bladder cancer unless the cancer is clinically stable and not requiring active treatment
11. Not have received chemotherapy or radiotherapy in the prior 30 days

Exclusion Criteria:

1. Immunosuppressed state (e.g. HIV, use of chronic steroids)
2. Fixed disease (clinical T4)
3. Active, uncontrolled infections
4. Hepatic impairment (SGOT >3x ULN)
5. Unhealed wounds
6. Patients at risk of pregnancy who are unwilling or unable to take effective contraception before rapamycin therapy, during therapy, and for 12 weeks after discontinuation of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Tissue pharmacodynamic (PD) response to TORC1 inhibition | 30 days
  PD response defined by significant phospho rpS6 Kinase 1 (S6K1) inhibition (comparing post-treatment to baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Svatek, MD,MSCI, Principal Investigator — UT Health Science Center San Antonio
Locations (1):
- UT Health Science Center San Antonio, San Antonio, Texas, United States